CLINICAL TRIAL: NCT00188890
Title: Early Diagnosis of Mesothelioma and Lung Cancer Following Asbestos Exposure Using Low-dose Computed Tomography
Brief Title: Early Diagnosis of Lung Cancer and Mesothelioma in Prior Asbestos Workers
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: Asbestos Screening Study
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Lung Cancer; Mesothelioma
Keywords: Lung Cancer; Mesothelioma; Asbestos; Screening; Early Diagnosis
MeSH Terms: conditions — Lung Neoplasms; Mesothelioma; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: prior occupational exposure at least 20 years ago to ASBESTOS and / or documented pleural plaques on a chest x-ray Must be 30 years of age or older. NO prior cancers, except non-melanic skin cancers

SUMMARY:
Occupational exposure to asbestos is known increase the risk of developing cancer of the lungs (bronchogenic carcinoma) or of the pleura (mesothelioma). Symptoms are subtle and non-specific, diagnosis is often late and the prognosis consequently is dismal. Currently there is no accepted non-invasive tool for the early diagnosis of mesothelioma or lung cancer in asbestos-exposed subjects. In the last decade, low-dose computed tomography (LDCT) has been successfully developed and validated for the early diagnosis of lung cancer in high-risk smokers. Malignant mesothelioma might, in an early stage, resemble a benign pleural plaque, which is a common finding after asbestos exposure. We target to develop low-dose CT as a tool to serially image the pleural plaques, quantify their individual and overall volume, compute the growth rate with time, and, as such, identify the presence of mesothelioma early, before symptoms occur.

DETAILED DESCRIPTION:
Background and Purpose:

Asbestos exposure may result in several different diseases to the lung and to the lining of the lung, the so-called pleura. Mostly they are benign, but there are two common malignant diseases in people with prior asbestos exposure, the so-called mesothelioma - which originates from the pleura - and cancer of the lung. Symptoms of any of these malignant diseases generally do not appear for 10-35 years after the first asbestos exposure, and include shortness of breath, chronic or new cough, coughing of blood, chest pain or weight loss. Unfortunately, these symptoms are most often causes by very advanced diseases, when patients can no longer be cured. Currently there is no accepted tool for the early diagnosis of mesothelioma or lung cancer in asbestos-exposed subjects available. Standard of care includes regular chest radiographs, which are not sufficient to show mesothelioma or lung cancer in an early stage.

A screening CT examination, also called CAT scan, of the lungs will be performed without intravenous contrast. The CT examination as such is not an experimental procedure, CAT scans are performed routinely since decades. However, in this particular case, this albeit standard examination is performed for the purposes of research only, it is not part of standard of care. The screening CT examination of the lungs takes less than 10-20 minutes to perform.

If no abnormalities are found on the initial examinations, you will be examined with one repeat screening CT of the chest after one year.

If pleural plaques or a nodule in the lungs is seen on your baseline CT, this will lead to further testing. Quite likely (approximately 1 in 3 chance), you will be invited for a follow-up CT 3 or 6 months. Further investigations will be chosen according to standard of care and will be explained to you at the time. These will be coordinated by your physician with Dr. Marc de Perrot, Department of Thoracic Surgery.

Secondly, there is evidence in other types of cancers such as cancers of the prostate and ovary, that analysis of blood may reveal protein markers that indicate the presence of cancer in the body. A companion blood analysis study is being undertaken in an effort to discover such markers for lung cancer and mesothelioma, so that the accuracy of CT-scan diagnosis for lung cancer may be further improved.

Both at the time of your baseline screening CT and at your annual follow-up screening CT, you will be asked to provide 5 ml (approximately 2 teaspoons full) blood sample through a needle stick. A blood-taking technician employed by the University Health Network or a certified nurse will carry out this procedure. Purpose of this study is to search in the blood for so-called "markers", substances in the blood which indicate that there is a cancer in the lungs or pleura.

Most of these markers are still in development, thus your blood will be stored and analyzed at a future date.

ELIGIBILITY:
Inclusion Criteria:

prior asbestos exposure at least 20 years ago and/or documented pleural plaques (chest x-ray evidence)

Resident of Ontario, Canada

Exclusion Criteria:

prior cancer (except non-melanotic skin cancer)

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: prior exposure to asbestos and or documented pleural plaques
Sampling Method: Non-Probability Sample
Enrollment: 1452 (Actual)
Dates: Start 2005-03 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2019-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Demetris Patsios, MD, Principal Investigator — University Health Network, Toronto; Marc de Perrot, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided